CLINICAL TRIAL: NCT00203099
Title: A Pilot, Multicenter, Open-label, One-group Study to Explore the Efficacy, Tolerability and Safety of the Combination of Glatiramer Acetate (GA) and N-Acetylcysteine (NAC) in Subjects With Relapsing Remitting Multiple Sclerosis (RR-MS)
Brief Title: Safety and Efficacy Study of Copaxone Administered in Combination With N-Acetylcysteine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA 9015
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Relapse Remitting Multiple Sclerosis
MeSH Terms: interventions — Glatiramer Acetate; Acetylcysteine

ARMS (1):
- Glatiramer Acetate, N-Acetylcysteine (Active Comparator)
  Interventions: Drug: Glatiramer Acetate, N-Acetylcysteine

INTERVENTIONS:
Drug: Glatiramer Acetate, N-Acetylcysteine — Subcutaneous glatiramer acetate 20 mg and concomitant oral administration of N-Acetylcysteine divided into two 2.5 g doses.

SUMMARY:
This study evaluates the effect of the therapy combining GA and NAC on disease activity as reflected by MRI parameters while assessing tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically Definite Multiple Sclerosis (CDMS) as defined by Poser et al (Ann Neurol 1983).
2. Subjects must have at least one T1 Gd-enhancing lesion in one of the pre-treatment MRI scans.
3. Subjects must have a relapsing-remitting disease course.
4. Subjects must have had at least one documented relapse within the last year prior to the screening visit (week -10).
5. Subjects must be relapse-free and not have taken corticosteroids (IV, IM and/or PO) within the 30 days prior to the screening visit.
6. Subjects may be male or female. Women of child- bearing potential must practice a medically acceptable method of birth control. Acceptable methods include oral contraceptive or double-barrier method (condom or IUD with spermicide).
7. Subjects must be between the ages of 18 and 50 years inclusive.
8. Subjects must be ambulatory, with a Kurtzke EDSS score of between 0 and 5.0 inclusive.
9. Subjects must be willing and able to give written informed consent prior to entering the study.

Exclusion Criteria:

1. Previous use of injected glatiramer acetate.
2. Previous use of cladribine within 2 years prior to screening visit (week -10).
3. Previous use of immunosuppressive agents in the last 6 months.
4. Use of experimental or investigational drugs, including I.V. immunoglobulin, within 6 months prior to study entry.
5. Use of interferon agents within 60 days prior to the screening visit.
6. Chronic corticosteroid (IV, IM and/or PO) treatment (more than 30 consecutive days) in the 6 months prior to study entry.
7. Chronic use of antioxidant substance(s), including NAC, (more than 30 consecutive days) within 60 days prior to the screening visit.
8. Previous total body irradiation or total lymphoid irradiation (TLI).
9. Pregnancy or breastfeeding.
10. Significant medical or psychiatric condition that affects the subject's ability to give informed consent, or to complete the study, or any condition which the investigator feels may interfere with participation in the study (e.g. alcohol or drug abuse).
11. A known history of uncontrolled asthma.
12. A known history of sensitivity to mannitol or acetylcysteine.
13. Inability to successfully undergo MRI scanning.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in the sum of T1 Gd-enhancing lesions as reflected by MRI | 46 weeks
  Change in the sum of T1 Gd-enhancing lesions measured at pre-treatment (weeks -10 [screening], -6 and 0 [baseline]) to the sum of T1 Gd-enhancing lesions measured in the last study trimester (weeks 28, 32 and 36 [termination]).

SECONDARY OUTCOMES:
MRI parameters | 46 Weeks
  Evaluation of secondary efficacy MRI parameters and assessments of tolerability and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Godin, MD, Study Director — Teva Neuroscience Canada